CLINICAL TRIAL: NCT00678002
Title: Quality of Life and Vulnerability in Pediatric Solid Organ Transplant Recipients
Brief Title: Quality of Life in Pediatric Transplant Patients
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Stacee Lerret, Advanced Practice Nurse, Medical College of Wisconsin
Other Study IDs: CHW 08/157; GC173
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Kidney Transplantation; Liver Transplantation; Heart Transplantation
Keywords: solid organ transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- QOL###: All child subjects in this cohort will be listed for or already have received a solid organ transplant (kidney, heart, or liver).

SUMMARY:
The goal of this study is to compare parent and child perceptions of wellness and vulnerability in children who have undergone solid organ transplant. It is hypothesized that there will be significant differences between parent and child perceptions.

DETAILED DESCRIPTION:
There are numerous studies that report on the quality of life in solid organ transplant recipients. However, very few studies target quality of life parameters for these children and their families across all solid organ transplantation. Furthermore, no literature directly addresses a comparison of perceptions and wellness, impact on family, and vulnerability in a comparative format by these distinct, but definitely related populations.

The goal of this study is to compare parent and child perceptions of wellness and vulnerability in children who have undergone solid organ transplant. It is hypothesized that there will be significant differences between parent and child perceptions. Outcomes will be measured by using five different instruments:

1. Pediatric Quality of Life Inventory (PedsQL)
2. PedsQL Family Impact Module
3. PedsQL Family Information Form
4. Functional Status II-R
5. Child Vulnerability Scale (CVS)

Patients will be enrolled at the time of transplant listing, or after transplant. Patients and families will complete the survey once every 6 months while the patient is active on the respective transplant waiting list. After transplant, the patients and families will be asked to complete the survey once every 6 months for the first two years and annually thereafter.

This study may provide us with an improved understanding of parent and child perceptions in wellness, impact on family, and vulnerability within each transplant group. The results may also indicate trend differences between these three populations. These differences may help to provide insight into family perspectives allowing for greater anticipatory guidance and targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* between newborn and 21 years old
* parent/child pairs of patients listed for or who have received a liver transplant, kidney transplant, or heart transplant

Exclusion Criteria:

* unwilling or unable to participate
* not in one of the above transplant groups
* non-English speaking

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children's Hospital of Wisconsin in the Hepatology Clinic, Cardiology Clinic, and Kidney Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2008-10; Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory | every 6 months

SECONDARY OUTCOMES:
Peds QL Family Impact Module | every 6 months
Peds QL Family Information Form | every 6 months
Functional Status II-R | every 6 months
Child Vulnerability Scale | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, CPNP, Principal Investigator — Medical College of Wisconsin; Gail Stendahl, CPNP, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Cole CR, Bucuvalas JC, Hornung RW, Krug S, Ryckman FC, Atherton H, Alonso MP, Balistreri WF, Kotagal U. Impact of liver transplantation on HRQOL in children less than 5 years old. Pediatr Transplant. 2004 Jun;8(3):222-7. doi: 10.1111/j.1399-3046.2004.00126.x. PMID 15176957
- [Background] Forsyth BW, Horwitz SM, Leventhal JM, Burger J, Leaf PJ. The child vulnerability scale: an instrument to measure parental perceptions of child vulnerability. J Pediatr Psychol. 1996 Feb;21(1):89-101. doi: 10.1093/jpepsy/21.1.89. PMID 8820075
- [Background] Freier MC, Babikian T, Pivonka J, Burley Aaen T, Gardner JM, Baum M, Bailey LL, Chinnock RE. A longitudinal perspective on neurodevelopmental outcome after infant cardiac transplantation. J Heart Lung Transplant. 2004 Jul;23(7):857-64. doi: 10.1016/j.healun.2003.08.003. PMID 15261181
- [Background] Goldstein SL, Graham N, Burwinkle T, Warady B, Farrah R, Varni JW. Health-related quality of life in pediatric patients with ESRD. Pediatr Nephrol. 2006 Jun;21(6):846-50. doi: 10.1007/s00467-006-0081-y. Epub 2006 Apr 20. PMID 16703376
- [Background] Green A, McSweeney J, Ainley K, Bryant J. In my shoes: children's quality of life after heart transplantation. Prog Transplant. 2007 Sep;17(3):199-207; quiz 208. doi: 10.1177/152692480701700307. PMID 17944159
- [Background] Manificat S, Dazord A, Cochat P, Morin D, Plainguet F, Debray D. Quality of life of children and adolescents after kidney or liver transplantation: child, parents and caregiver's point of view. Pediatr Transplant. 2003 Jun;7(3):228-35. doi: 10.1034/j.1399-3046.2003.00065.x. PMID 12756049
- [Background] Mussatto K, Tweddell J. Quality of life following surgery for congenital cardiac malformations in neonates and infants. Cardiol Young. 2005 Feb;15 Suppl 1:174-8. doi: 10.1017/s1047951105001253. No abstract available. PMID 15934713
- [Background] Pollock-BarZiv SM, Anthony SJ, Niedra R, Dipchand AI, West LJ. Quality of life and function following cardiac transplantation in adolescents. Transplant Proc. 2003 Nov;35(7):2468-70. doi: 10.1016/j.transproceed.2003.08.028. PMID 14611988
- [Background] Roy, C., & Andrews, H. A. (1991). The roy adaptation model: The definitive statement. East Norwalk, Connecticut: Prentice Hall.
- [Background] Schulz KH, Wein C, Boeck A, Rogiers X, Burdelski M. Cognitive performance of children who have undergone liver transplantation. Transplantation. 2003 Apr 27;75(8):1236-40. doi: 10.1097/01.TP.0000062843.10397.32. PMID 12717209
- [Background] Stuber ML. Psychiatric aspects of organ transplantation in children and adolescents. Psychosomatics. 1993 Sep-Oct;34(5):379-87. doi: 10.1016/S0033-3182(93)71840-X. PMID 8140186
- [Background] Sweet SC, Wong HH, Webber SA, Horslen S, Guidinger MK, Fine RN, Magee JC. Pediatric transplantation in the United States, 1995-2004. Am J Transplant. 2006;6(5 Pt 2):1132-52. doi: 10.1111/j.1600-6143.2006.01271.x. PMID 16613592
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Wray J, Radley-Smith R. Depression in pediatric patients before and 1 year after heart or heart-lung transplantation. J Heart Lung Transplant. 2004 Sep;23(9):1103-10. doi: 10.1016/j.healun.2003.08.018. PMID 15454178
- [Background] Wray J, Radley-Smith R. Longitudinal assessment of psychological functioning in children after heart or heart-lung transplantation. J Heart Lung Transplant. 2006 Mar;25(3):345-52. doi: 10.1016/j.healun.2005.09.018. Epub 2006 Jan 18. PMID 16507430
- [Background] Wray J, Radley-Smith R. Beyond the first year after pediatric heart or heart-lung transplantation: Changes in cognitive function and behaviour. Pediatr Transplant. 2005 Apr;9(2):170-7. doi: 10.1111/j.1399-3046.2005.00265.x. PMID 15787788